CLINICAL TRIAL: NCT00154739
Title: A Phase II Randomized Trial of Gemcitabine/Cisplatin Versus Gemcitabine/Epirubicin in Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Gemcitabine/Cisplatin Versus Gemcitabine/Epirubicin for Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 46S1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2008-08-04 (Estimated); Status verified 2005-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Combination, Chemotherapy,non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin; Epirubicin

INTERVENTIONS:
Drug: Gemcitabine
Drug: Cisplatin
Drug: Epirubicin

SUMMARY:
The purpose of this study is to evaluate the efficacy of gemcitabine/cisplatin versus gemcitabine/epirubicin in Stage IIIB/IV NSCLC in terms of response rate and overall survival.

DETAILED DESCRIPTION:
Most patients suffered from nausea, vomiting and prolonged anorexia after cisplatin treatment. Epirubicin is an anthracycline that was used widely in the treatment of cancer. Our previous study of an epirubicin and paclitaxel combination in non-small cell lung cancer patients showed a response rate of 52.6% and good median survival. However, most patients suffered from paclitaxel-related neurotoxicity.

Chemotherapy may increase an average of 1 to 2 months of median survival in inoperable non-small cell lung cancer patients treated with chemotherapy. However, chemotherapy may not provide a cure for these patients. Reduction of side effects and enhancement of life quality of the patients are as important as life prolongation for these patients. We designed a combination chemotherapy using gemcitabine with epirubicin in the treatment of inoperable non-small cell lung cancer. The treatment will be compared to gemcitabine and cisplatin combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of stage IIIB/IV NSCLC
* No prior chemotherapy
* Age > 18 years
* ECOG score < 0 to 2
* Bi-dimensionally measurable lesions
* WBC > 4,000/ml, ANC > 1,500/ml, platelets>100,000/ml
* Hb>10g/dl.
* ALT/AST < 5 times x UNL, bilirubin < 1.5times x UNL, creatinine < 1.25 times x UNL, normal calcium level
* Life expectancy > 12 weeks

Exclusion Criteria:

* CNS metastases, Concomitant myelosuppressive radiotherapy, C/T, hormonal therapy or immunotherapy.
* Active congestive heart failure, angina and/or arrhythmia requiring therapy or previous myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 1998-10; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to explore efficacy of gemcitabine and epirubicin in the treatment of NSCLC patients who need palliative chemotherapy.

SECONDARY OUTCOMES:
The secondary objective of this study is to compare efficacy (response rate，overall survival) of gemcitabine/epirubicin to gemcitabine/cisplatin in the treatment of inoperable NSCLC.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hsin Yang, M.D., Ph.D., Principal Investigator — Department of Oncology, National Taiwan University Hospital; Ann-Lii Cheng, M.D., Ph.D., Study Chair — Department of Oncology, National Taiwan University Hospital
Locations (1):
- Department of Oncology, National Taiwan University Hospital, Taipei, Taiwan